CLINICAL TRIAL: NCT06913764
Title: First- or Second- Class Compression Hosiery After Endovenous Laser With Sclerotherapy and Ambulatory Phlebectomy: Randomized Controlled Trial (FISCHER)
Brief Title: First- or Second- Class Compression Hosiery After Endovenous Laser With Sclerotherapy and Ambulatory Phlebectomy
Acronym: FISCHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow City Hospital named after A.K. Eramishantsev (Other Government)
Collaborators: Pirogov Russian National Research Medical University (Other); Vishnevsky Center of Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1/2025
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Varicose Veins; Chronic Venous Disorder; Chronic Venous Insufficiency (CVI); Venous Reflux; Great Saphenous Vein (GSV) With Venous Reflux Disease
Keywords: Varicose veins; Varicose disease; Compression therapy; medical compression stockings; MCS; venous disease; veins; vein surgery; elastic hosiery; compression hosiery; endovenous laser; endovenous laser ablation; thermal ablation; sclerotherapy; microsclerotherapy; phlebectomy; ambulatory phlebectomy; elastic compression
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Intervention Model Description: A single-center, open, non-inferiority randomized controlled trial with a blinded outcome assessor
Who Masked: Outcomes Assessor
Masking Description: A single-center, open, non-inferiority randomized controlled trial with a blinded outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Class 1 (18-21 mm Hg at the ankle level) above-knee graduated compression stockings (Experimental): All participants will undergo measurement of the affected limb at standard points to select the appropriate size of compression stockings. Then, the clinical class of chronic venous disease will be assessed for the study participants according to the CEAP classification, the severity of chronic venous disease will be evaluated using the VCSS scale, quality of life will be measured using the CIVIQ-20 questionnaire, and the intensity of venous-specific symptoms will be assessed using a numerical rating scale. After the surgical intervention, a class 1 compression stocking will be put on, which they will wear continuously for 24 hours; thereafter, it must be worn during the daytime for 28 days. Upon discharge, patients will receive a diary in which they will record postoperative pain and the fact of wearing the compression garment each day for 14 days. Follow-up visits will be scheduled for 14 days and 28 days after the surgical intervention.
  Interventions: Device: class I compression stockings of the RAL-GZ 387 standard: 1 month using
- Class 2 (23-32 mm Hg at the ankle level) above-knee graduated compression stockings (Active Comparator): All participants will undergo measurement of the affected limb at standard points to select the appropriate size of compression stockings. Then, the clinical class of chronic venous disease will be assessed for the study participants according to the CEAP classification, the severity of chronic venous disease will be evaluated using the VCSS scale, quality of life will be measured using the CIVIQ-20 questionnaire, and the intensity of venous-specific symptoms will be assessed using a numerical rating scale. After the surgical intervention, a class 2 compression stocking will be put on, which they will wear continuously for 24 hours; thereafter, it must be worn during the daytime for 28 days. Upon discharge, patients will receive a diary in which they will record postoperative pain and the fact of wearing the compression garment each day for 14 days. Follow-up visits will be scheduled for 14 days and 28 days after the surgical intervention.
  Interventions: Device: class II compression stockings of the RAL-GZ 387 standard: 1 month using

INTERVENTIONS:
Device: class I compression stockings of the RAL-GZ 387 standard: 1 month using — Class 1 (RAL-GZ 387 standard: 18-21 mm Hg at the ankle level) above-knee graduated compression stockings
  Arms: Class 1 (18-21 mm Hg at the ankle level) above-knee graduated compression stockings
Device: class II compression stockings of the RAL-GZ 387 standard: 1 month using — Class 2 (RAL-GZ 387 standard: 23-32 mm Hg at the ankle level) above-knee graduated compression stockings
  Arms: Class 2 (23-32 mm Hg at the ankle level) above-knee graduated compression stockings

SUMMARY:
Investigators hypothesize that first class compression therapy during the postoperative period will improve patient adherence due to easier application and reduced discomfort. Therefore, planning to compare the effectiveness of fist class versus second class compression therapy two weeks after EVLA of the great saphenous vein with concomitant combined sclerotherapy and ambulatory phlebectomy of tributaries.

DETAILED DESCRIPTION:
In recent decades, significant advancements have emerged in varicose vein treatment. Endovenous laser ablation (EVLA) and radiofrequency ablation (RFA) have become the leading techniques for eliminating trunk reflux, while microfoam sclerotherapy and ambulatory phlebectomy are most commonly used for treating tributaries. Post-intervention, patients typically receive recommendations to wear second-class compression stockings to reduce postoperative pain, ecchymosis, and hematomas. However, the optimal duration, regimen, and compression class remain poorly defined. Meanwhile, a growing surgical community advocates for eliminating compression therapy during the postoperative period altogether, citing low patient compliance rates (15-74%). The primary factors driving non-compliance include discomfort while wearing hosiery and difficulties with donning and doffing, suggesting compression hosiery characteristics may significantly impact adherence. Recent meta-analyses support compression therapy's benefits, demonstrating reduced postoperative pain levels and faster return to normal activities among patients using postoperative compression. Additionally, both national and international clinical guidelines recommend compression therapy for at least one week following thermal ablations. Investigators hypothesize that first class compression therapy during the postoperative period will improve patient adherence due to easier application and reduced discomfort. Therefore, planning to compare the effectiveness of first class versus second class compression therapy two weeks after EVLA of the great saphenous vein with concomitant combined sclerotherapy and ambulatory phlebectomy of tributaries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Varicose veins of the lower extremities (CEAP classification C2-C5)
* Varicose disease in the great saphenous vein (GSV) and its tributaries
* Planned endovenous laser ablation of the GSV trunk with concomitant combined sclerotherapy and phlebectomy of tributaries
* Technical success of intervention (complete ablation of the GSV)
* Signed informed consent for study participation

Exclusion Criteria:

* Primary reflux outside the GSV trunk
* History of or acute deep vein thrombosis
* Deep vein insufficiency
* GSV recanalization post-intervention
* Clinical class C6 of chronic venous disease (CVD) according to CEAP classification
* Contraindications or limitations for prolonged compression therapy, including but not limited to chronic arterial diseases of the lower extremities (any severity), skin diseases
* Pathological conditions of lower limbs causing non-venous pain
* Use of vasoactive medications within 1 month before/after surgery
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Level of postoperative pain at 14 days | 14 days
  The intensity of postoperative pain is subjectively assessed by the patient on a 10-centimeter numeric scale daily. The range is from 0 (no pain) to 10 (pain of maximal intensity).

SECONDARY OUTCOMES:
Area (centimeter square) of ecchymosis | 14 days
  Assessed by an expert by measuring ecchymoses using a specialized smartphone application "LesionMeter".
Number of patients with clinical manifestations of phlebitis at 14 days | 14 days
  Clinical significant appearance of signs of inflammation (hyperemia, swelling, pain) of the superficial veins
The change of clinical class of chronic venous disease according to the CEAP classification in the operated lower limb at 28 days | 28 days
  The class of chronic venous disease in the operated lower limb is assessed by an expert during a clinical examination based on the CEAP classification.
VCSS score at 14 days | 14 days
  The severity of chronic venous disease (CVD) in the target lower limb is assessed during clinical examination using the updated Venous Clinical Severity Score (VCSS). Ranges from 0 to 30. The maximal score indicates more severe CVD.
VCSS score at 28 days | 28 days
  The severity of chronic venous disease (CVD) in the target lower limb is assessed during clinical examination using the updated Venous Clinical Severity Score (VCSS). Ranges from 0 to 30. The maximal score indicates more severe CVD.
The intensity of primary venous-specific symptoms on the operated lower limb according to a numerical rating scale at 14 days | 14 days
  Venous-specific symptoms are assessed by the patient independently using a numerical rating scale. The range is from 0 to 100, with a minimum score indicating the best quality of life.
The intensity of primary venous-specific symptoms on the operated lower limb according to a numerical rating scale at 28 days | 28 days
  Venous-specific symptoms are assessed by the patient independently using a numerical rating scale. The range is from 0 to 100, with a minimum score indicating the best quality of life.
CIVIQ-20 score at 14 days | 14 days
  The quality of life is assessed by the patient independently according to the vein-specific questionnaire Chronic Lower Limb Venous Insufficiency Questionnaire - 20 items (CIVIQ-20). range 0-100, a minimal score indicates the best quality of life.
CIVIQ-20 score at 28 days | 28 days
  The quality of life is assessed by the patient independently according to the vein-specific questionnaire Chronic Lower Limb Venous Insufficiency Questionnaire - 20 items (CIVIQ-20). range 0-100, a minimal score indicates the best quality of life.
Compliance with the use of Medical Compression Stockings (MCS) | 14 days
  Compliance with the use of MCS is assessed based on the study of the patient's diaries in Groups 1 and 2 as a proportion of the number of days when the patient used MCS for at least 8 hours to the total duration of prescribed compression (14 days), represented as a percentage (n[MCS]/14*100%). It ranges from 0% (no compliance) to 100% (absolute compliance).
Comfort with the use of MCS at 14 days | 14 days
  The patients subjectively assess their comfort when using MCS using a 100-cm numeric rating scale, which ranges from 0 (no comfort) to 10 (absolute comfort).
Comfort with the use of MCS at 28 days | 28 days
  The patients subjectively assess their comfort when using MCS using a 100-cm numeric rating scale, which ranges from 0 (no comfort) to 10 (absolute comfort).
Difficulty in putting on a compression stocking at 14 days | 14 days
  Patients subjectively assess the level of difficulty in putting on the compression stockings using a 100-point numerical scale, which ranges from 0 (no difficulty) to 100 (absolute difficulty).
Difficulty in putting on a compression stocking at 28 days | 28 days
  Patients subjectively assess the level of difficulty in putting on the compression stockings using a 100-point numerical scale, which ranges from 0 (no difficulty) to 100 (absolute difficulty).
The circumference length of the narrowest part of the calf above the ankle one month after the intervention at 28 days | 28 days
  The circumference length of the narrowest part of the calf was measured by an expert using a measuring tape.

CONTACTS AND LOCATIONS:
Overall Officials: Hovsep P. Manjikian, MD, Study Chair — Moscow City Hospital named after A.K. Eramishantsev; Boris Danelian, MD, Principal Investigator — Moscow City Hospital named after A.K. Eramishantsev; Hovsep Manjikyan, MD, Principal Investigator — Moscow City Hospital named after A.K. Eramishantsev
Locations (1):
- Moscow City Hospital named after A.K. Eramishantsev, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Local regulations

REFERENCES:
- [Background] Rabe E, Partsch H, Hafner J, Lattimer C, Mosti G, Neumann M, Urbanek T, Huebner M, Gaillard S, Carpentier P. Indications for medical compression stockings in venous and lymphatic disorders: An evidence-based consensus statement. Phlebology. 2018 Apr;33(3):163-184. doi: 10.1177/0268355516689631. Epub 2017 Feb 22. PMID 28549402
- [Background] Ma F, Xu H, Zhang J, Premaratne S, Gao H, Guo X, Yang T. Compression Therapy Following Endovenous Thermal Ablation of Varicose Veins: A Systematic Review and Meta-Analysis. Ann Vasc Surg. 2022 Mar;80:302-312. doi: 10.1016/j.avsg.2021.09.035. Epub 2021 Nov 11. PMID 34774690
- [Background] Hu H, Wang J, Wu Z, Liu Y, Ma Y, Zhao J. No Benefit of Wearing Compression Stockings after Endovenous Thermal Ablation of Varicose Veins: A Systematic Review and Meta-Analysis. Eur J Vasc Endovasc Surg. 2022 Jan;63(1):103-111. doi: 10.1016/j.ejvs.2021.09.034. Epub 2021 Nov 11. PMID 34776296
- [Background] Reich-Schupke S, Murmann F, Altmeyer P, Stucker M. Quality of life and patients' view of compression therapy. Int Angiol. 2009 Oct;28(5):385-93. PMID 19935593
- [Background] Kankam HKN, Lim CS, Fiorentino F, Davies AH, Gohel MS. A Summation Analysis of Compliance and Complications of Compression Hosiery for Patients with Chronic Venous Disease or Post-thrombotic Syndrome. Eur J Vasc Endovasc Surg. 2018 Mar;55(3):406-416. doi: 10.1016/j.ejvs.2017.11.025. Epub 2018 Jan 9. PMID 29329662
- [Background] Ayala A, Guerra JD, Ulloa JH, Kabnick L. Compliance with compression therapy in primary chronic venous disease: Results from a tropical country. Phlebology. 2019 May;34(4):272-277. doi: 10.1177/0268355518798153. Epub 2018 Sep 6. PMID 30189813
- [Background] Raju S, Hollis K, Neglen P. Use of compression stockings in chronic venous disease: patient compliance and efficacy. Ann Vasc Surg. 2007 Nov;21(6):790-5. doi: 10.1016/j.avsg.2007.07.014. PMID 17980798
- [Background] Nicolaides A, Kakkos S, Baekgaard N, Comerota A, de Maeseneer M, Eklof B, Giannoukas AD, Lugli M, Maleti O, Myers K, Nelzen O, Partsch H, Perrin M. Management of chronic venous disorders of the lower limbs. Guidelines According to Scientific Evidence. Part I. Int Angiol. 2018 Jun;37(3):181-254. doi: 10.23736/S0392-9590.18.03999-8. No abstract available. PMID 29871479
- [Background] Gianesini S, Obi A, Onida S, Baccellieri D, Bissacco D, Borsuk D, Campisi C, Campisi CC, Cavezzi A, Chi YW, Chunga J, Corda D, Crippa A, Davies A, De Maeseneer M, Diaz J, Ferreira J, Gasparis A, Intriago E, Jawien A, Jindal R, Kabnick L, Latorre A, Lee BB, Liew NC, Lurie F, Meissner M, Menegatti E, Molteni M, Morrison N, Mosti G, Narayanan S, Pannier F, Parsi K, Partsch H, Rabe E, Raffetto J, Raymond-Martimbeau P, Rockson S, Rosukhovski D, Santiago FR, Schul A, Schul M, Shaydakov E, Sibilla MG, Tessari L, Tomaselli F, Urbanek T, van Rijn MJ, Wakefield T, Wittens C, Zamboni P, Bottini O. Global guidelines trends and controversies in lower limb venous and lymphatic disease: Narrative literature revision and experts' opinions following the vWINter international meeting in Phlebology, Lymphology & Aesthetics, 23-25 January 2019. Phlebology. 2019 Sep;34(1 Suppl):4-66. doi: 10.1177/0268355519870690. No abstract available. PMID 31495256
- [Background] Lurie F, Lal BK, Antignani PL, Blebea J, Bush R, Caprini J, Davies A, Forrestal M, Jacobowitz G, Kalodiki E, Killewich L, Lohr J, Ma H, Mosti G, Partsch H, Rooke T, Wakefield T. Compression therapy after invasive treatment of superficial veins of the lower extremities: Clinical practice guidelines of the American Venous Forum, Society for Vascular Surgery, American College of Phlebology, Society for Vascular Medicine, and International Union of Phlebology. J Vasc Surg Venous Lymphat Disord. 2019 Jan;7(1):17-28. doi: 10.1016/j.jvsv.2018.10.002. PMID 30554745
- [Background] Kolluri R, Hays KU, Gohel MS. Foam Sclerotherapy Augmented Phlebectomy (SAP) Procedure for Varicose Veins: Report of a Novel Technique. EJVES Short Rep. 2018 Nov 16;41:16-18. doi: 10.1016/j.ejvssr.2018.10.007. eCollection 2018. PMID 30519649
- [Background] Carradice D, Mekako AI, Hatfield J, Chetter IC. Randomized clinical trial of concomitant or sequential phlebectomy after endovenous laser therapy for varicose veins. Br J Surg. 2009 Apr;96(4):369-75. doi: 10.1002/bjs.6556. PMID 19283745
- [Background] De Maeseneer MG, Kakkos SK, Aherne T, Baekgaard N, Black S, Blomgren L, Giannoukas A, Gohel M, de Graaf R, Hamel-Desnos C, Jawien A, Jaworucka-Kaczorowska A, Lattimer CR, Mosti G, Noppeney T, van Rijn MJ, Stansby G, Esvs Guidelines Committee, Kolh P, Bastos Goncalves F, Chakfe N, Coscas R, de Borst GJ, Dias NV, Hinchliffe RJ, Koncar IB, Lindholt JS, Trimarchi S, Tulamo R, Twine CP, Vermassen F, Wanhainen A, Document Reviewers, Bjorck M, Labropoulos N, Lurie F, Mansilha A, Nyamekye IK, Ramirez Ortega M, Ulloa JH, Urbanek T, van Rij AM, Vuylsteke ME. Editor's Choice - European Society for Vascular Surgery (ESVS) 2022 Clinical Practice Guidelines on the Management of Chronic Venous Disease of the Lower Limbs. Eur J Vasc Endovasc Surg. 2022 Feb;63(2):184-267. doi: 10.1016/j.ejvs.2021.12.024. Epub 2022 Jan 11. No abstract available. PMID 35027279
- [Background] Gloviczki P, Lawrence PF, Wasan SM, Meissner MH, Almeida J, Brown KR, Bush RL, Di Iorio M, Fish J, Fukaya E, Gloviczki ML, Hingorani A, Jayaraj A, Kolluri R, Murad MH, Obi AT, Ozsvath KJ, Singh MJ, Vayuvegula S, Welch HJ. The 2023 Society for Vascular Surgery, American Venous Forum, and American Vein and Lymphatic Society clinical practice guidelines for the management of varicose veins of the lower extremities. Part II: Endorsed by the Society of Interventional Radiology and the Society for Vascular Medicine. J Vasc Surg Venous Lymphat Disord. 2024 Jan;12(1):101670. doi: 10.1016/j.jvsv.2023.08.011. Epub 2023 Aug 29. PMID 37652254
- [Background] Kamaev AA, Bulatov VL, Vakhratyan PE, Volkov AM, Volkov AS, Gavrilov EK, Golovina VI, Efremova OI, Ivanov OO, Ilyukhin EA, Katorkin SE, Konchugova TV, Kravtsov PF, Maksimov SV, Mzhavanadze ND, Pikhanova ZhM, Pryadko SI, Smirnov AA, Sushkov SA, Chabbarov RG, Shimanko AI, Yakushkin SN, Apkhanova TV, Derkachev SN, Zolotukhin IA, Kalinin RE, Kirienko AI, Kulchitskaya DB, Pelevin AV, Petrikov AS, Rachin AP, Seliverstov EI, Stoyko YuM, Suchkov IA. Clinical Guidelines. Varicose Veins. Flebologiya. 2022;16(1):41-108. (In Russ.). https://doi.org/10.17116/flebo20221601141
- [Background] Luebke T, Brunkwall J. Systematic review and meta-analysis of endovenous radiofrequency obliteration, endovenous laser therapy, and foam sclerotherapy for primary varicosis. J Cardiovasc Surg (Torino). 2008 Apr;49(2):213-33. PMID 18431342
- [Background] Darwood RJ, Theivacumar N, Dellagrammaticas D, Mavor AI, Gough MJ. Randomized clinical trial comparing endovenous laser ablation with surgery for the treatment of primary great saphenous varicose veins. Br J Surg. 2008 Mar;95(3):294-301. doi: 10.1002/bjs.6101. PMID 18278775
- See also: Related Info — https://gkbe.ru